CLINICAL TRIAL: NCT00311168
Title: Reduce Ventricular Pacing Using Ventricular Intrinsic Preference: VIP™ Study
Brief Title: Reduction of Right Ventricular Pacing Using the Feature Ventricular Intrinsic Preference (VIP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CRD343
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Results first posted 2021-07-19 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia | interventions — Methods; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- VIP On, Then VIP Off (Experimental): Participants first have VIP programmed On after randomization until 3 months, followed by VIP programmed Off from 3 to 6 months.
  Interventions: Device: Intervention/treatment
- VIP Off, Then VIP On (Experimental): Participants first have VIP programmed Off after randomization until 3 months, followed by VIP programmed On from 3 to 6 months.
  Interventions: Device: Intervention/treatment

INTERVENTIONS:
Device: Intervention/treatment — Device: VIP On
  Device: VIP Off

SUMMARY:
The purpose of this study is to evaluate the efficacy of the VIP™ feature (available in dual chamber Victory® devices) to reduce unnecessary RV pacing, and to determine if patients with implanted SJM pacemakers will benefit by using VIP™ rather than only a programmed AV/PV delay.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been implanted with dual chamber SJM Victory® device with VIP™ for 1 month (± 2 weeks).
* At the time of pacemaker implant, VIP™ is programmed "OFF".
* At the time of enrollment, patient is paced in the RV ≤ 60% of the time.
* Patient is medically stable.

Exclusion Criteria:

* Patient has evidence of complete AV block, such that ventricular pacing would be required as part of the patient's routine management.
* Patient is indicated for AF Suppression.
* Patient has persistent or chronic atrial fibrillation.
* Patient is unable to comply with the follow-up visits due to geographical, psychological, or any other reasons.
* Patient is currently participating in another device research study.
* Patient is younger than 18 years of age.
* Patient is pregnant.
* Patients life expectancy is less than 12 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clay Cohorn, Study Director — Abbott
Locations (1):
- Abbott, Sylmar, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 134 of 135 subjects were randomized. One subject was not randomized.
Groups:
- VIP On, Then VIP Off: Participants first have the VIP algorithm programmed On after randomization until 3 months, followed by VIP programmed Off from 3 to 6 months.
  Intervention/treatment:
  Device: VIP On Device: VIP Off
- VIP Off, Then VIP On: Participants first have VIP programmed Off after randomization until 3 months, followed by VIP programmed On from 3 to 6 months.
  Intervention/treatment:
  Device: VIP Off Device: VIP On
Period: First Intervention
Arm/Group | VIP On, Then VIP Off | VIP Off, Then VIP On
Started | 66 | 68
Completed | 59 | 62
Not Completed | 7 | 6
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Other | 2 | 2
Period: Second Intervention
Arm/Group | VIP On, Then VIP Off | VIP Off, Then VIP On
Started | 59 | 62
Completed | 49 | 58
Not Completed | 10 | 4
Not completed — Lost to Follow-up | 9 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: A total of 135 subjects were enrolled in the study and 134 of these 135 subjects were randomized. The 134 randomized subjects are included in the baseline analysis population.
Groups:
- VIP On, Then VIP Off: Participants first have VIP programmed On after randomization until 3 months, followed by VIP programmed Off from 3 to 6 months.
  Intervention/treatment:
  Device: VIP On Device: VIP Off
- VIP Off, Then VIP On: Participants first have VIP programmed Off after randomization until 3 months, followed by VIP programmed On from 3 to 6 months.
  Intervention/treatment:
  Device: VIP On Device: VIP Off
- Total: Total of all reporting groups
Arm/Group | VIP On, Then VIP Off | VIP Off, Then VIP On | Total
Number analyzed (Participants) | 66 | 68 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (16.1) | 75.6 (10.4) | 74.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 67/68 subjects (VIP On, then VIP Off) and 64/66 subjects (VIP Off, then VIP On) have gender information collected on the CRF
  Participants
    number analyzed (Participants) | 64 | 67 | 131
    Female | 30 | 37 | 67
    Male | 34 | 30 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Intrinsic Ventricular Events
Description: This outcome measured evaluated the difference in the percentage of intrinsic ventricular events between VIP On and VIP Off. A higher percentage indicates more intrinsic ventricular events and a lower amount of unnecessary RV pacing.
Time Frame: 6 months after randomization
Population: The analysis population includes patients enrolled in the study with data available on the outcome measure at 6 months after randomization.
Measure: Mean (Standard Deviation); unit: % of intrinsic ventricular events
Groups:
- VIP On: VIP On Group
  * VIP On, then VIP Off
  * VIP Off, then VIP On
- VIP Off: VIP Off Group
  * VIP On, then VIP Off
  * VIP Off, then VIP On
Arm/Group | VIP On | VIP Off
Number analyzed (Participants) | 107 | 107
% of intrinsic ventricular events | 82.7 (28.5) | 22.8 (31.3)
Statistical Analysis 1: Comparison: VIP On vs VIP Off; Test type: Superiority — A target of an 80% reduction in percentage of ventricular pacing with VIP™ is proposed in this study. In order to achieve an 80% power of detecting an 80% reduction in the percentage of ventricular paced events and using a two group two-sided t-test of equal means, a minimum sample size of 39 patients per group was required. To account for possible withdrawal or loss to follow-up, this study targeted to enroll 100 patients (50 per group); p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -60.2, 95% CI 2-sided [-67.5 to -52.9], Standard Deviation 19 — Mean difference in the percentage of intrinsic ventricular events is presented as, VIP Off - VIP On

2. Secondary Outcome: Incidence of Arrhythmias
Description: This outcome measure evaluated the difference in the percentage of time a patient spent in atrial tachycardia/atrial fibrillation (arrhythmia burden) calculated by the device between VIP On and VIP Off.
Time Frame: 6 months after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of burden
Arm/Group | VIP On | VIP Off
Number analyzed (Participants) | 102 | 102
percentage of burden | 3.6 (13) | 2 (6.3)

3. Secondary Outcome: Percentage of Atrial Sensing to Ventricular Sensing (%PR)
Description: This outcome measure evaluated the difference in the percentage of atrial sensing to ventricular sensing (%PR) detected by the device between VIP On and VIP Off. A higher percentage indicates more intrinsic ventricular events and a lower amount of unnecessary RV pacing.
Time Frame: 6 months after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PR
Arm/Group | VIP On | VIP Off
Number analyzed (Participants) | 107 | 107
percentage of PR | 41.9 (34.2) | 12.3 (21)

4. Secondary Outcome: Percentage of Atrial Sensing to Ventricular Pacing (%PV)
Description: This outcome measure evaluated the difference in the percentage of Atrial Sensing to Ventricular Pacing (%PV) between VIP On and VIP Off. A lower percentage indicates more intrinsic ventricular events and a lower amount of unnecessary RV pacing.
Time Frame: 6 months after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PV
Arm/Group | VIP On | VIP Off
Number analyzed (Participants) | 108 | 108
percentage of PV | 8.3 (18.7) | 37.4 (37)

5. Secondary Outcome: Percentage of Atrial Pacing to Ventricular Sensing (%AR)
Description: This outcome measure evaluated the difference in the percentage of Atrial Pacing to Ventricular Sensing (%AR) between VIP On and VIP Off. A higher percentage indicates more intrinsic ventricular events and a lower amount of unnecessary RV pacing.
Time Frame: 6 months after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of AR
Arm/Group | VIP On | VIP Off
Number analyzed (Participants) | 108 | 108
percentage of AR | 40.5 (35) | 10.4 (20.3)

6. Secondary Outcome: Percentage of Atrial Pacing to Ventricular Pacing (%AV)
Description: This outcome measure evaluated the difference in the percentage of Atrial Pacing to Ventricular Pacing (%AV) between VIP On and VIP Off. A lower percentage indicates more intrinsic ventricular events and a lower amount of unnecessary RV pacing.
Time Frame: 6 months after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of AV
Arm/Group | VIP On | VIP Off
Number analyzed (Participants) | 107 | 107
percentage of AV | 10.5 (21.6) | 38.1 (35.2)

7. Secondary Outcome: Percentage of Patients Experiencing a Study-Related Adverse Event
Description: This outcome measure evaluated the incidence of study-related adverse events between VIP On and VIP Off.
Time Frame: 6 months after randomization
Measure: Count of Participants; unit: Participants
Groups:
- VIP On: VIP On Period
- VIP Off: VIP Off Period
Arm/Group | VIP On | VIP Off
Number analyzed (Participants) | 134 | 134
Participants | 0 | 2

8. Secondary Outcome: Number of Auto Mode Switch Events
Description: This outcome measure evaluated the difference in the number of auto mode switch events between VIP On and VIP Off.
Time Frame: 6 months after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | VIP On | VIP Off
Number analyzed (Participants) | 104 | 104
Counts | 3.1 (11.6) | 1.9 (5.9)

ADVERSE EVENTS:
Time Frame: 6 months for each intervention
Description: Safety Population included all subjects who were randomized and received at least one of the interventions (VIP On or VIP Off).
Arm/Group | VIP On | VIP Off
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/134
Serious Adverse Events (participants affected / at risk) | 0/134 | 1/134
Other Adverse Events (participants affected / at risk) | 0/134 | 1/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIP On (N=134) | VIP Off (N=134)
LEAD DISLODGEMENT OR MIGRATION (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIP On (N=134) | VIP Off (N=134)
DIMINISHING R-WAVE AMPLITUDE (Product Issues) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No